CLINICAL TRIAL: NCT02910674
Title: Dario Blood Glucose Monitoring System - Android Devices User Performance
Brief Title: Dario Blood Glucose Monitoring System - Android Devices User Performance Study Report
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LabStyle Innovations Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CP-0004
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Results first posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

ARMS (1):
- One Arm (Other): This is a comparative diagnostic study, no interventional actions are being taken.
  Interventions: Device: Dario Blood Glucose Monitoring System

INTERVENTIONS:
Device: Dario Blood Glucose Monitoring System — Accuracy with usability assessment

SUMMARY:
The purpose of this study is to evaluate the accuracy of the Dario Blood Glucose Monitoring System as compared to a reference method (Yellow Springs Instrument 2300 STAT Plus) and to evaluate the usability of the device when used by laypersons.

DETAILED DESCRIPTION:
The objectives for this study are to evaluate the blood glucose level results obtained from the subject's fingertip using the Dario Blood Glucose Monitoring System paired with a reference device from one of three Android smart mobile device families as compared to the results from the Yellow Springs Instrument 2300 STAT Plus. The usability of the Dario Blood Glucose Monitoring System when paired with a reference device from one of three Android smart mobile device families and used by laypersons is also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subject has Type 1 or Type II diabetes
* Subject speaks and reads English proficiently
* Subject is able and agrees to sign the informed consent form (minor subjects must be accompanied by a parent or legal guardian to provide consent for their participation in the study)

Exclusion Criteria:

* Subject has medical training or works in the field of blood glucose monitoring systems.
* Subject is critically ill.
* Subject has an impairment that prevents him/her from following the study procedures.
* Subject has any condition that the Principal Investigator believes may interfere in the subject's participation in the study.
* Hematocrit levels outside the range of 20%-60%.

Ages: 13 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-07; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Barbara Davis Center, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Diabetes (Type I or II), Ages 13-80: Males and females with diabetes (type I or II), ages 13-80 recruited through advertisement, outpatient clinics, physician offices, and similar sources.
Period: Overall Study
Arm/Group | Diabetes (Type I or II), Ages 13-80
Started | 102
Completed | 102
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diabetes (Type I or II), Ages 13-80
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 6
  Black or African American | 1
  White | 90
  More than one race | 4
  Unknown or Not Reported | 0
Subjects with Type I and Type II diabetes [Count of Participants; unit: Participants] | 102

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Glucose Concentrations (%)
Description: Accuracy acceptability is defined as follows:
  Ninety-five percent (95%) of the individual glucose results shall fall within +/-15 mg/dL of the results of the Dario's measurement at glucose concentrations < 75 mg/dL and within +/- 20% at glucose concentrations greater than or equal to 75 mg/dL.
  The accuracy of the Dario Blood Glucose Monitoring System when used with Android operating system smart mobile devices was assessed against the Yellow Springs Instrument 2300 STAT Plus.
Time Frame: 1 Day
Measure: Number (95% Confidence Interval); unit: percentage of measurements within range
Arm/Group | Diabetes (Type I or II), Ages 13-80
Number analyzed (Participants) | 102
percentage of measurements within range | 97.4 [95 to 100]

2. Primary Outcome: Average Rank of the Indication of "How Would Rate Your Success in Operating Dario BGMS"
Description: Using a scale of 1-5 where 1-completely fails, 2-unsuccessful, 3-Partially successful, 4-successful, 5-very successful.
  Average rank of 3.5 ('average'/'successful') or above in question #2 - How would you rate your success in operating Dario™ BGMS?
Time Frame: 1 Day
Population: 102 ranked their success in operating Dario™ BGMS 1-5. 1- Completely failed, 5- Very successful
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | One Arm
Number analyzed (Participants) | 102
score on a scale | 4.4 [1 to 5]

3. Primary Outcome: Average Rank of the Indication of "How Easy Was it to Operate the Dario™ BGMS on the First Time?"
Description: Using a scale of 1-5 where 1-very hard, 2-hard, 3-average, 4-easy, 5-very easy.
  An average rank of 3 ('average') or above in question #3 - How easy was it to operate the Dario™ BGMS on the first time?
Time Frame: 1 Day
Population: 102 ranked their ease in operating Dario™ BGMS 1-5. 1- Very Hard, 5- Very Easy
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | One Arm
Number analyzed (Participants) | 102
score on a scale | 3.9 [1 to 5]

4. Primary Outcome: Percent of Participants Responding 'YES' on the Question "Did You Successfully Obtain Measurement Result Using the Dario™ BGMS?"
Description: The acceptance criteria for this question is: at least ninety percent (90%) need to answer 'Yes' on question #1 - Did you successfully obtain measurement result using the Dario™ BGMS?
  100% of subjects (102 of 102) answered "Yes" to this question.
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | One Arm
Number analyzed (Participants) | 102
Participants | 102

ADVERSE EVENTS:
Time Frame: 4 Days
Description: Reporting requirements are provided in compliance with 21 CFR 812.150(b) (1). All-Cause Mortality: No mortalities were recorded during the study Serious Adverse Events: No serious adverse events were recorded during the study Other (Not Including Serious) Adverse Events: No other adverse events were recorded during the study
Arm/Group | Diabetes (Type I or II), Ages 13-80
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes